CLINICAL TRIAL: NCT05432375
Title: A Phase 1 Study to Investigate the Safety, Pharmacokinetics, and Efficacy of Tinostamustine, a Novel Alkylating and Deacetylase Inhibiting Molecule, as Adjuvant Treatment in Patients With Newly Diagnosed Unmethylated MGMT-promoter Glioblastoma
Brief Title: Study of Tinostamustine for Adjuvant Treatment of Glioblastoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mundipharma Research Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EDO S101-1006
Record Dates: First submitted 2022-06-09; First posted 2022-06-27 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — tinostamustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tinostamustine (Experimental): Infusion delivered over 60 minutes
  Interventions: Drug: Tinostamustine

INTERVENTIONS:
Drug: Tinostamustine — infusion given over 60 minutes

SUMMARY:
The study is designed as an open label, multi-center, Phase 1 study of single agent tinostamustine, used as adjuvant treatment in patients with newly diagnosed GBM who are MGMT unmethylated and have completed concomitant treatment with temozolomide and radiation. Treatment with adjuvant tinostamustine will start within 5 weeks of completion of concomitant temozolomide and radiation. The study is designed to define the MTD by evaluating toxicities during dose escalation. Tinostamustine will be administered on Day 1 of a 21-day treatment cycle.

The total number of treatment cycles is 12 for patients who continue to benefit from treatment without disease progression or intolerable toxicity. Patients will enter a "3+3" design with dose escalation/de-escalation depending on safety from the last treated cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have Grade 4 isocitrate dehydrogenase (IDH) wild type GBM with local pathology confirmed MGMT-promoter unmethylated status.
2. Patients must have undergone surgical resection of the GBM tumour and have completed standard radiation therapy with concurrent temozolomide and must not have clear signs of progression such as new disease outside the radiation area, neurological progression, or clinical progression that leads to other exclusion criteria.
3. A baseline brain magnetic resonance imaging (MRI) obtained no more than 14 days prior to first dose of tinostamustine on a stable or decreasing dose of steroids for at least 5 days, is required prior to entrance of a patient onto the study.
4. Patients must be registered on the study within 5 weeks of completion of concurrent chemoradiation.
5. Patient must be willing and able to provide written informed consent for the study.
6. Age ≥18 years on day of signing informed consent.
7. Prescribed treatment with concomitant temozolomide must be consistent with the EORTC-22981-26981 study (NCT00006353). The dose must be 75 mg/m2 daily for the 6 to 6.5 weeks of radiation therapy. The patient must have completed at least 75% of temozolomide dosing during radiotherapy.
8. Confirmed IDH wild type. The presence of an IDH mutation will be exclusionary for study enrolment. IDH mutation testing by at least one method (such as immunohistochemistry for IDH1 R132H) must be performed as part of standard of care and no mutation must be found (i.e., IDH wild type). If a mutation is identified, then the patient will be ineligible.
9. Patients must have a performance status of ≥60 on the Karnofsky Performance Scale (KPS).
10. If patient is on steroids, patient must be on a stable or decreasing dose of steroids for at least 5 days at the time of baseline brain MRI.
11. Demonstrate adequate organ function as defined in Table 3. All screening laboratories should be performed within 14 days (+/- 2 days) of treatment initiation.
12. Serum potassium and magnesium at least at the lowest limit of normal (LLN) range, before every tinostamustine administration. If it is below LLN, supplementation is permissible.
13. Female patients of childbearing potential should have a negative serum pregnancy test within 48 hours of starting first dose of tinostamustine.
14. Female study participants of childbearing potential and their partners, and male study participants who intend to be sexually active with a woman of childbearing potential, must be willing to use at least TWO highly effective forms of contraception. This should start from the time of study enrolment and continue throughout tinostamustine administration. Female study participants of childbearing potential must continue using contraception for at least 6 months after the last administration of the tinostamustine. Female study participants should be willing to have a pregnancy test performed at screening, on Day -1 of each tinostamustine administration and at tinostamustine discontinuation. Male study participants who are sexually active with a woman of childbearing potential should also use a condom during treatment and for at least 90 days after the last administration of tinostamustine. Vasectomised males are considered fertile; therefore, vasectomised partners and patients must be willing to use a secondary method of effective birth control. Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the tinostamustine. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the patient.

Exclusion Criteria:

1. Patient has received prior interstitial brachytherapy, implanted chemotherapy, or therapeutics delivered by local injection or convection enhanced delivery. Prior treatment with Gliadel® wafers will be excluded. Concomitant use of the tumour treating fields will also be excluded.
2. Use of chemotherapy or immunotherapy within 21 days (apart from TMZ), use of targeted therapy within 14 days or 5 times the half-life of the agent, whichever is longer, prior to the first dose of tinostamustine. After the respective durations mentioned above, patients may be enrolled if they have recovered from any related toxicities ≥ Grade 1 (except alopecia). This applies to any prior systemic anticancer therapy including investigational agents.
3. Any serious medical condition that interferes with adherence to study procedures.
4. Patient has had prior chemotherapy (excluding radiotherapy + temozolomide), targeted small molecule therapy, within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤Grade 1 at baseline) from AEs due to a previously administered agent.

   1. Note: Patients with ≤Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   2. Note: If patients received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
5. Patients with a history of a second malignancy diagnosed within 3 years of study enrolment or have a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
6. Implanted pacemaker or implantable cardiac defibrillator or New York Heart Association (NYHA) Stage III/IV congestive heart failure or with the following arrhythmias: atrial fibrillation/flutter with poor rate control; documented sustained ventricular tachycardia (defined as >30 seconds or requiring cardioversion before 30 seconds have elapsed) or TdP; ventricular pre excitation (Wolff Parkinson White syndrome) Brugada Syndrome; complete left bundle branch block (LBBB); QRS >120 ms; myocardial infarction or acute coronary syndrome within previous 6 months.
7. Severe chronic obstructive pulmonary disease (COPD) or severe uncontrollable hypertension.
8. Patients who did not complete at least 75% of temozolomide dosing during radiotherapy per EORTC-22981-26981 study.
9. Patients who had a platelet count <75,000/mm3 during concomitant temozolomide therapy during radiation.
10. Patients with QTc interval (Fridericia's formula) >450 ms.
11. Patients who are on treatment with drugs known to prolong the QT/QTc interval. Selective serotonin reuptake inhibitors (SSRIs): Patients treated with a SSRI AND displaying a QTc prolongation are NOT eligible in the study.

    Nevertheless, there is no need to stop or change a SSRI if a patient is on a stable dose AND with no impact on QT/QTc interval, since it is not expected that plasma concentration of the SSRI will be affected by the administration of tinostamustine.
12. Patient has known gliomatosis cerebri, leptomeningeal disease, extracranial disease, or multifocal disease. Patient has multifocal GBM, defined as discrete sites of contrast enhancing disease without contiguous T2/FLAIR abnormality that require distinct radiotherapy ports. Satellite lesions that are associated with a contiguous area of T2/FLAIR abnormality as the main lesion(s) and that are encompassed within the same radiotherapy port as the main lesion(s) are permitted.
13. Patient has an active infection requiring systemic therapy.
14. Patient has an ongoing or previous history of spontaneous intratumoral haemorrhage.
15. Patient has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator.
16. Patient has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
17. Patient is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit.
18. Patient has a known history of human immunodeficiency virus (HIV type 1 or 2 antibodies). Testing not required.
19. Patient has known active hepatitis B (e.g., HBs Ag reactive) or hepatitis C (e.g., HCV RNA [qualitative]) is detected.
20. Patient has received a live vaccine within 30 days prior to the first dose of tinostamustine.
21. Contraindication for undergoing MRIs.
22. Use of any drug with histone deacetylase (HDAC) inhibiting activity including use of valproate in any of its indications (epilepsy, mood disorder). Valproate, due to its HDAC inhibiting activity is contraindicated. For those patients on valproate, valproate will need to be discontinued and switched to a different anti epileptic agent or psychotropic agent. A washout period of 4 days from valproate acid will be allowed prior to enrolling into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-11-10 (Actual); Study Completion 2024-11-10 (Actual)

PRIMARY OUTCOMES:
Dose Limiting toxicity | cycle 1 of treatment. Cycle 1 is 21 days duration with infusion given on day 1
  Toxicity will be evaluated according to the most current version of the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) toxicity criteria

SECONDARY OUTCOMES:
Anti-tumour activity | Approx 1 year from start of treatment
  Response assessment in neuro-oncology (RANO) criteria (to assess mPFS, PFS, ORR, OS, duration of response [DoR])
Pharmacokinetic assessment | cycle 1 of treatment. Cycle is 21 days duration with infusion given on day 1
  plasma concentrations of tinostamustine

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Janik, MD, Study Director — Mundipharma Research Limited
Locations (5):
- Spain (3):
  - Hospital Universitario Vall d'Hebron, Barcelona, Spain, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid, Spain, Madrid
  - South Texas Accelerated Research Therapeutics (START), Madrid
- Switzerland (2):
  - Kantonsspital, Sankt Gallen
  - University Hospital, Zurich

IPD SHARING:
Plan to Share IPD: No